CLINICAL TRIAL: NCT00494390
Title: Neuartige Kontaktlose Biometrische Messungen
Brief Title: Evaluation Study for a Non-Contact Biometer
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Haag-Streit AG (Industry)
Other Study IDs: kek-98/07; Insel 1351
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2007-07

CONDITIONS: Cataract; Pseudophakia; Myopia; Hyperopia; Aphakia
Keywords: Biometry; corneal opacity; astigmatism; refraction
MeSH Terms: conditions — Cataract; Pseudophakia; Myopia; Hyperopia; Aphakia; Corneal Opacity; Astigmatism

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether a new non-contact biometer, is as accurate as the the available gold-standard.

DETAILED DESCRIPTION:
The features of a not yet commercial available new biometer will be compared to available contact and non contact biometers in different patient groups.

ELIGIBILITY:
Inclusion Criteria:

1. 18 year or older
2. Normal eye
3. Cataract
4. Corneal abnormality (scar, opacity, transplant)
5. refractive corneal surgery
6. Pseudophakia
7. Aphakia
8. Silicon oil
9. refractive IOL

2.-9. (at least one yes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Goldblum, MD, Principal Investigator — www.insel.ch
Locations (1):
- Department of Ophthalmology, University Hospital, Bern, Switzerland